CLINICAL TRIAL: NCT04089410
Title: Direct and Cross Effects of Adaptation to Systemic Hyperthermia: Impact on Quality of Life, Neurohormonal and Psychophysiological Human Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dudnik Elena Nikolaevna, Associate professor, I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: АААА-А19-119012190093-4
Record Dates: First submitted 2019-09-06; First posted 2019-09-13 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Hypoxia, Altitude; Exercise Tolerance; Metabolic Disturbance; Quality of Life
Keywords: Adaptation; Systemic hyperthermia; Quality of life; Neuro-visceral interactions; Preventive medical technologies; Personalized approach; Neuroplasticity; Brain derived neurotrophic factor; Irisin; Heat Shock proteins
MeSH Terms: conditions — Altitude Sickness | interventions — Restraint, Physical; Standing Position; Psychological Tests

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperthermic Fitness Treatment (Active Comparator): Participants will fill out study questionnaires. After basic body measurements subjects will undergo the HFT.
  Interventions: Device: Hyperthermic Fitness Treatment (HFT); Other: Physical Examination; Other: Assessment of Cardiorespiratory Fitness; Other: Autonomic Balance, Orthostatic and Hypoxic tolerance; Other: Psychological Testing; Other: Measurement of Blood Markers
- Attenuated heating (Placebo Comparator): Participants will fill out study questionnaires. After basic body measurements subjects will undergo the placebo-HFT.
  Interventions: Device: Placebo Hyperthermic Fitness Treatment; Other: Physical Examination; Other: Assessment of Cardiorespiratory Fitness; Other: Autonomic Balance, Orthostatic and Hypoxic tolerance; Other: Psychological Testing; Other: Measurement of Blood Markers

INTERVENTIONS:
Device: Hyperthermic Fitness Treatment (HFT) — The Hyperthermic Fitness Treatment uses Alfa Basic capsule, an ergonomic camera in which a participant may take a lying position and undergo hyperthermia procedures (infrared heating with intracapsule temperature increase up to 80 degrees C◦), the head being outside the camera blown by cool air with a built-in ventilator. HFT is comparable to dry sauna bathing. Core body temperatures will be raised to 37.5-38.5°C◦. Recommended duration of one HFT session is 40 min. All the HFT group participants while undergoing sessions in the Cocoon will be dressed in bathing suits.
  Arms: Hyperthermic Fitness Treatment
Device: Placebo Hyperthermic Fitness Treatment — Attenuated heating with less heat set (20-30 degrees C◦). This results in no increase of core body temperature. The participant will still feel heat and will see similar lighting and hear similar sounds as those occurring during actual HFT, and will be in the capsule for the same period of time.
  Arms: Attenuated heating
Other: Physical Examination — Resting hearth rate (HR), Systolic and Diastolic blood pressure (SBP and DBP) values are measured twice in supine position using an automatic tonometer after 5 min of rest.
  Body mass (BM) and height are measured to calculate Body Mass Index. Body composition is assessed with the use of portable body-impedance-meter for the whole body impedance-analysis.
  Body core temperature, Blood pressure (BP) and Heart rate (HR) are measured before and right after each session. Arterial oxygen saturation (SpO2) and HR is monitored continuously by the use of a pulse oximeter, attached to the index fingertip of non dominant hand.
Other: Assessment of Cardiorespiratory Fitness — An assessment of exercise tolerance and cardiorespiratory fitness (ET, CRF) is carried out with the use of Cardiopulmonary Exercise Test - CPET). Testing is carried out using a gas analyzer and an Intertrack treadmill. Evaluation of gas exchange parameters conducted according to a given program - Cardiopulmonary load testing.
Other: Autonomic Balance, Orthostatic and Hypoxic tolerance — 1. Evaluation of Autonomic balance is assesed using Heart Rate Variability (HRV) analysis. The HRV test relies on a 5-min RR interval (time in milliseconds between two R waves of the electrocardiogram complex) recorded at rest for 5 min supine (SU) followed of 5 min resting time. Measurement of the interval duration between two R waves of the cardiac electrical activity are performed with a HR monitor.
  2. Orthostatic tolerance is assessed after ANS balance assessment by HRV analysis to continue RR intervals registration for 3 min after participant was asked to stand up taking a vertical position near the couch.
  3. The individual sensitivity to hypoxia is determined by conducting a 10-minute hypoxic test (HT) - breathing through a facial mask by a gas mixture with 11% of O2, with minute-by-minute monitoring of HR and hemoglobin saturation by oxygen (SaO2). Arterial blood pressure is recorded before and after HT.
Other: Psychological Testing — 1. Medical Outcomes Study Short-Form 36-Item Health Survey (SF-36), which is a self-completed quantity of health-related QoL.
  2. Participants are asked to complete the Pittsburgh Sleep Quality Index (PSQI), a retrospective self-report measure assessing their quality of sleep during the last three weeks preceding the study.
  3. Anxiety level is estimated by using State and Trait Anxiety Scales (SA and TA) developed by Ch. Spielberger
  4. Subjective Ratings of Thermosensation and Pain.Participants rate their comfort, thermosensation, and pain by fixing results in visual-analogous scale (VAS) while passing each of HFT treatment.
Other: Measurement of Blood Markers — Periferal venous blood (10 ml) sumples of the fastest (overnight fast) study subjects are withdrawn by a qualified laboratory technician via aseptic technique from the antecubital vein in the sitting position, using sterile needles and are collected. Serum BDNF, HGH, HSPs (60, 70, 90) concentrations are determined.

SUMMARY:
Life expectancy and quality of human life are important indicator of the sustainable development of the society. At the same time, the physical, functional, emotional and psychological components of the of the quality of life evaluation are subjected to be evaluated objectively and corrected using modern medical and socio-psychological methods. According to a fair number of experts, the arsenal of means for functional rehabilitation and health promotion is limited, and its expansion is only possible on the basis of the principles of adaptation medicine and their translation from experimental research into specific preventive and health-promoting technologies.

The study is aimed at the development in molecular-endocrine, neuro-visceral and psychophysiological complex mechanisms of human long-term adaptation to systemic modern heating device-based hyperthermia for the development of medical technology focused on optimization in physical functioning, neuro-autonomic regulation, psycho-emotional status and stress- resistance as objective characteristics of humans' quality of life in working age.

The novelty of the project is the disclosure of key mechanisms of adaptational direct and cross-effects to the prolonged systemic individually dosed hyperthermia underlying the optimization of stress-resistance, psycho-physiological status and exercise tolerance of practically healthy persons and leading to an increase in the subjectively perceived quality of life.

The discovery of the mechanisms of hyperthermically induced neuroplasticity (in terms of the dynamics of oxidative stress, heat shock proteins and the brain derived neurotrophic factor) will also have a scientific significance, which in the long term prospectives may play a role in the development of technics for the prevention and rehabilitation of age-associated neuro-degenerative processes and diseases.

DETAILED DESCRIPTION:
Hyperthermic Fitness Treatment (HFT) is proved in many applied and clinical trials to be a helpful tool for enhancing thermal acclimation, physical tolerance and endurance, improving cardiovascular dysfunctions, normalizing metabolic status and body weight in patients with chronic non-infectious diseases and in aged healthy individuals. Clinical effects of hyperthermia acclimation or repeated sauna's sessions were investigated in series of well-designed placebo-controlled studies at different cohorts of Bronchial Asthma (BA), Chronic Obstructive Pulmonary Disease (COPD), Cardiovascular Disease (CVD) Metabolic Syndrome and Obesity (MS-O) patients, qualified professional sportsmen and healthy volunteers.

Effects of sauna bathing and hyperthermic treatments (acclimation to systemic, whole body dosed hyperthermia, which leads to core temperature increase on 2,0-2,5oC) are accurately described in well-controlled medical studies, performed by experienced researchers imposing different protocols (from 1 session lasting 15-20 min, daily 1 week up to 2 sessions per day, 3 weeks).

The generalized result of the most trials suggests adaptation to hyperthermia (sauna bathing sessions) is accompanied by a multi-faceted molecular, cellular, organic and systemic, organismic responses - by progressively increased resistance to thermal stressors, increased bronchial conductivity and pulmonary ventilation, sweating; stimulated activation of neuro-humoral and cardiovascular systems, boosted microcirculation and, as a consequence, providing more efficient transport and utilization of O2 by body tissues, resulting in increase of exercise tolerance, physical activity, normalization of appetite, balancing thermogenesis and heat release.

Mechanisms underlying the described clinical effects are partially connected with increased production of some neurotransmitters, hormones and peptides, among them - Brain derived neurotropic factor (BDNF), Somatotropin (Human Growth Hormone - HGH), Heat Shock Proteins family as cell signaling pathways inducers etc.

In spite of difference in study design, protocols, and hyperthermic mashines - devices, it is safe to make the conclusion that periodic individually adapted hyperthermic sessions are capable to induce haematological, neuro-humoral, cardiorespiratory and antioxidant adaptation to provide pathogenetic treatment and rehabilitation of patients with chronic non-infectious diseases.

Enhanced stress resistance and improved oxygen transfer/utilization are basic mechanisms whereby the organism increases its resistance to any physical and environmental stressors and to variety of pathogenic factors.

The described Hyperthermic Fitness Treatment (HFT) method is safe, has no significant complications or adverse side effects and is generally very well tolerated by sportsmen, healthy persons and different clinical patients' groups.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, young healthy volunteers
* Age > 19 years (20 - 30)
* Gender: male
* Healthy state (no chronic noninfectious diseases, documented by medical check-up results, obtained in 1-2 months before, not later), mobility (absence of orthopedic problems), satisfactory level of fitness
* Ability to perform activities of daily living
* Ability to attend all treatments and clinical-laboratory measurements
* Signed informed consent form

Exclusion Criteria:

* Infectious diseases
* Increased body temperature before any step of the study
* Individual hyperthermia (sauna) intolerance
* Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the volunteer to participate in this study e.g. expected survival <1 year
* Participation in another clinical study with an investigational product within 28 days prior to enrolment or previous randomization to an investigational product in another ongoing clinical study

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Change in Cardiopulmonary Exercise Test | Week 1
  An assessment of exercise tolerance and cardiorespiratory fitness (ET, CRF) is carried out by Cardiopulmonary Exercise Test - CPET) with the use of Fitmate MED gas analyzer (COSMED, Italy) and an Intertrack treadmill (Shiller, Switzerland).
Change in Cardiopulmonary Exercise Test | Week 5
  An assessment of exercise tolerance and cardiorespiratory fitness (ET, CRF) is carried out by Cardiopulmonary Exercise Test - CPET) with the use of Fitmate MED gas analyzer (COSMED, Italy) and an Intertrack treadmill (Shiller, Switzerland).
Change in Cardiopulmonary Exercise Test | Week 13
  An assessment of exercise tolerance and cardiorespiratory fitness (ET, CRF) is carried out by Cardiopulmonary Exercise Test - CPET) with the use of Fitmate MED gas analyzer (COSMED, Italy) and an Intertrack treadmill (Shiller, Switzerland).
Measurement of Blood Markers | Week 1
  Serum BDNF, HGH, HSPs (60, 70, 90), Irisin concentrations
Measurement of Blood Markers | Week 5
  Serum BDNF, HGH, HSPs (60, 70, 90), Irisin concentrations
Measurement of Blood Markers | Week 13
  Serum BDNF, HGH, HSPs (60, 70, 90), Irisin concentrations
Psychological stress tolerance: Quality of Life | Week 1
  We assessed QoL using the Medical Outcomes Study Short-Form 36-Item Health Survey (SF-36), which is a self-completed quantity of health-related QoL. This questionnaire comprises eight domains covering physical functioning, vitality, role-physical, social functioning, bodily pain, role-emotional, general health and mental health. A high score indicates a better QoL characteristic. Furthermore, there are two summary scores which summarize two domains: first the Mental Component Summary and second the Physical Component Summary.
Psychological stress tolerance: Quality of Life | Week 5
  We assessed QoL using the Medical Outcomes Study Short-Form 36-Item Health Survey (SF-36), which is a self-completed quantity of health-related QoL. This questionnaire comprises eight domains covering physical functioning, vitality, role-physical, social functioning, bodily pain, role-emotional, general health and mental health. A high score indicates a better QoL characteristic. Furthermore, there are two summary scores which summarize two domains: first the Mental Component Summary and second the Physical Component Summary.
Psychological stress tolerance: Quality of Life | Week 13
  We assessed QoL using the Medical Outcomes Study Short-Form 36-Item Health Survey (SF-36), which is a self-completed quantity of health-related QoL. This questionnaire comprises eight domains covering physical functioning, vitality, role-physical, social functioning, bodily pain, role-emotional, general health and mental health. A high score indicates a better QoL characteristic. Furthermore, there are two summary scores which summarize two domains: first the Mental Component Summary and second the Physical Component Summary.
Psychological stress tolerance: Sleep Quality | Week 1
  Assessment of Sleep Quality(The Pittsburgh Sleep Quality Index)
Psychological stress tolerance: Sleep Quality | Week 5
  Assessment of Sleep Quality(The Pittsburgh Sleep Quality Index)
Psychological stress tolerance: Sleep Quality | Week 13
  Assessment of Sleep Quality(The Pittsburgh Sleep Quality Index)
Psychological stress tolerance: Anxiety level | Week 1
  Assessment of Anxiety level (State and Trait Anxiety Scales developed by Ch. Spielberger)
Psychological stress tolerance: Anxiety level | Week 5
  Assessment of Anxiety level (State and Trait Anxiety Scales developed by Ch. Spielberger)
Psychological stress tolerance: Anxiety level | Week 13
  Assessment of Anxiety level (State and Trait Anxiety Scales developed by Ch. Spielberger)

SECONDARY OUTCOMES:
Hearth rate | Up to week 13
  Resting hearth rate (HR) values are measured twice in supine position.
Blood pressure | Up to week 13
  Systolic and Diastolic blood pressure (SBP and DBP) values are measured twice in supine position.
Body Mass Index | Change between baseline and week 13
  Body mass (BM) in kilograms and height in meters are measured (Seca 888 scale, Hamburg, Germany) to calculate Body Mass Index (BMI, in kg/m2). Metabolic rate at rest is measured in supine position by Fitmate MED gas analyzer (COSMED, Italy).
Metabolic rate | Change between baseline and week 13
  Metabolic rate at rest is measured in supine position by Fitmate MED gas analyzer (COSMED, Italy).
Body mass | Up to week 13
  Body mass is measured in kilograms
Height | 1 week
  Height is measured in meters
Autonomic Balance, Orthostatic and Hypoxic tolerance. | Change between baseline and week 13
  For the assessment of participants' autonomic regulation Heart Rate Variability (HRV) analysis is selected.Briefly, the HRV test relied on a 5-min RR interval (time in milliseconds between two R waves of the electrocardiogram complex) recorded at rest for 5 min supine (SU) followed of 5 min resting time. Measurement of the interval duration between two R waves of the cardiac electrical activity is performed with a HR monitor (VNS-Spectrum hardware and software complex (Neurosoft Company, Ivanovo, Russia).

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Glazachev, MD, Study Chair — Sechenov University
Locations (1):
- Students health and quality of life laboratory, Moscow, Russia

REFERENCES:
- [Background] Ansley L, Marvin G, Sharma A, Kendall MJ, Jones DA, Bridge MW. The effects of head cooling on endurance and neuroendocrine responses to exercise in warm conditions. Physiol Res. 2008;57(6):863-872. Epub 2007 Nov 30. PMID 18052690
- [Background] An JJ, Liao GY, Kinney CE, Sahibzada N, Xu B. Discrete BDNF Neurons in the Paraventricular Hypothalamus Control Feeding and Energy Expenditure. Cell Metab. 2015 Jul 7;22(1):175-88. doi: 10.1016/j.cmet.2015.05.008. Epub 2015 Jun 11. PMID 26073495
- [Background] Aspelund A, Antila S, Proulx ST, Karlsen TV, Karaman S, Detmar M, Wiig H, Alitalo K. A dural lymphatic vascular system that drains brain interstitial fluid and macromolecules. J Exp Med. 2015 Jun 29;212(7):991-9. doi: 10.1084/jem.20142290. Epub 2015 Jun 15. PMID 26077718
- [Background] Bath KG, Schilit A, Lee FS. Stress effects on BDNF expression: effects of age, sex, and form of stress. Neuroscience. 2013 Jun 3;239:149-56. doi: 10.1016/j.neuroscience.2013.01.074. Epub 2013 Feb 10. PMID 23402850
- [Background] Bekinschtein P, Cammarota M, Katche C, Slipczuk L, Rossato JI, Goldin A, Izquierdo I, Medina JH. BDNF is essential to promote persistence of long-term memory storage. Proc Natl Acad Sci U S A. 2008 Feb 19;105(7):2711-6. doi: 10.1073/pnas.0711863105. Epub 2008 Feb 8. PMID 18263738
- [Background] Bekinschtein P, Oomen CA, Saksida LM, Bussey TJ. Effects of environmental enrichment and voluntary exercise on neurogenesis, learning and memory, and pattern separation: BDNF as a critical variable? Semin Cell Dev Biol. 2011 Jul;22(5):536-42. doi: 10.1016/j.semcdb.2011.07.002. Epub 2011 Jul 7. PMID 21767656
- [Background] Biro S, Masuda A, Kihara T, Tei C. Clinical implications of thermal therapy in lifestyle-related diseases. Exp Biol Med (Maywood). 2003 Nov;228(10):1245-9. doi: 10.1177/153537020322801023. PMID 14610268
- [Background] Black EAE, Smith PM, McIsaac W, Ferguson AV. Brain-derived neurotrophic factor acts at neurons of the subfornical organ to influence cardiovascular function. Physiol Rep. 2018 May;6(10):e13704. doi: 10.14814/phy2.13704. PMID 29802680
- [Background] Buchheit M, Papelier Y, Laursen PB, Ahmaidi S. Noninvasive assessment of cardiac parasympathetic function: postexercise heart rate recovery or heart rate variability? Am J Physiol Heart Circ Physiol. 2007 Jul;293(1):H8-10. doi: 10.1152/ajpheart.00335.2007. Epub 2007 Mar 23. No abstract available. PMID 17384128
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cabanac M, Caputa M. Natural selective cooling of the human brain: evidence of its occurrence and magnitude. J Physiol. 1979 Jan;286:255-64. doi: 10.1113/jphysiol.1979.sp012617. PMID 439025
- [Background] Cacioppo JT, Berntson GG, Binkley PF, Quigley KS, Uchino BN, Fieldstone A. Autonomic cardiac control. II. Noninvasive indices and basal response as revealed by autonomic blockades. Psychophysiology. 1994 Nov;31(6):586-98. doi: 10.1111/j.1469-8986.1994.tb02351.x. PMID 7846219
- [Background] Carlino D, Francavilla R, Baj G, Kulak K, d'Adamo P, Ulivi S, Cappellani S, Gasparini P, Tongiorgi E. Brain-derived neurotrophic factor serum levels in genetically isolated populations: gender-specific association with anxiety disorder subtypes but not with anxiety levels or Val66Met polymorphism. PeerJ. 2015 Oct 29;3:e1252. doi: 10.7717/peerj.1252. eCollection 2015. PMID 26539329
- [Background] Cotman CW, Berchtold NC, Christie LA. Exercise builds brain health: key roles of growth factor cascades and inflammation. Trends Neurosci. 2007 Sep;30(9):464-72. doi: 10.1016/j.tins.2007.06.011. Epub 2007 Aug 31. PMID 17765329
- [Background] Edelmann E, Lessmann V, Brigadski T. Pre- and postsynaptic twists in BDNF secretion and action in synaptic plasticity. Neuropharmacology. 2014 Jan;76 Pt C:610-27. doi: 10.1016/j.neuropharm.2013.05.043. Epub 2013 Jun 18. PMID 23791959
- [Background] Enette L, Vogel T, Fanon JL, Lang PO. Effect of Interval and Continuous Aerobic Training on Basal Serum and Plasma Brain-Derived Neurotrophic Factor Values in Seniors: A Systematic Review of Intervention Studies. Rejuvenation Res. 2017 Dec;20(6):473-483. doi: 10.1089/rej.2016.1886. Epub 2017 Jun 28. PMID 28498065
- [Background] Ferris LT, Williams JS, Shen CL. The effect of acute exercise on serum brain-derived neurotrophic factor levels and cognitive function. Med Sci Sports Exerc. 2007 Apr;39(4):728-34. doi: 10.1249/mss.0b013e31802f04c7. PMID 17414812
- [Background] Ftaiti F, Jemni M, Kacem A, Zaouali MA, Tabka Z, Zbidi A, Grelot L. Effect of hyperthermia and physical activity on circulating growth hormone. Appl Physiol Nutr Metab. 2008 Oct;33(5):880-7. doi: 10.1139/H08-073. PMID 18923562
- [Background] Gibson OR, Taylor L, Watt PW, Maxwell NS. Cross-Adaptation: Heat and Cold Adaptation to Improve Physiological and Cellular Responses to Hypoxia. Sports Med. 2017 Sep;47(9):1751-1768. doi: 10.1007/s40279-017-0717-z. PMID 28389828
- [Background] Gibson OR, Tuttle JA, Watt PW, Maxwell NS, Taylor L. Hsp72 and Hsp90alpha mRNA transcription is characterised by large, sustained changes in core temperature during heat acclimation. Cell Stress Chaperones. 2016 Nov;21(6):1021-1035. doi: 10.1007/s12192-016-0726-0. Epub 2016 Aug 11. PMID 27511024
- [Background] Goekint M, Roelands B, Heyman E, Njemini R, Meeusen R. Influence of citalopram and environmental temperature on exercise-induced changes in BDNF. Neurosci Lett. 2011 Apr 25;494(2):150-4. doi: 10.1016/j.neulet.2011.03.001. Epub 2011 Mar 6. PMID 21385602
- [Background] Goldstein DS, Bentho O, Park MY, Sharabi Y. Low-frequency power of heart rate variability is not a measure of cardiac sympathetic tone but may be a measure of modulation of cardiac autonomic outflows by baroreflexes. Exp Physiol. 2011 Dec;96(12):1255-61. doi: 10.1113/expphysiol.2010.056259. Epub 2011 Sep 2. PMID 21890520
- [Background] Gryka D, Pilch W, Szarek M, Szygula Z, Tota L. The effect of sauna bathing on lipid profile in young, physically active, male subjects. Int J Occup Med Environ Health. 2014 Aug;27(4):608-18. doi: 10.2478/s13382-014-0281-9. Epub 2014 Jul 7. PMID 25001587
- [Background] Gupte AA, Bomhoff GL, Swerdlow RH, Geiger PC. Heat treatment improves glucose tolerance and prevents skeletal muscle insulin resistance in rats fed a high-fat diet. Diabetes. 2009 Mar;58(3):567-78. doi: 10.2337/db08-1070. Epub 2008 Dec 10. PMID 19073766
- [Background] Hannuksela ML, Ellahham S. Benefits and risks of sauna bathing. Am J Med. 2001 Feb 1;110(2):118-26. doi: 10.1016/s0002-9343(00)00671-9. PMID 11165553
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Iguchi M, Littmann AE, Chang SH, Wester LA, Knipper JS, Shields RK. Heat stress and cardiovascular, hormonal, and heat shock proteins in humans. J Athl Train. 2012 Mar-Apr;47(2):184-90. doi: 10.4085/1062-6050-47.2.184. PMID 22488284
- [Background] Iwase S, Kawahara Y, Nishimura N, Nishimura R, Miwa C, Kataoka Y, Kobayashi C, Suzuki T, Shigaraki M, Maeda Y, Takada H, Watanabe Y. A comparison of head-out mist bathing, with or without facial fanning, with head-out half-body low-water level bathing in humans--a pilot study. Int J Biometeorol. 2014 Jul;58(5):999-1005. doi: 10.1007/s00484-013-0685-4. Epub 2013 Jun 12. PMID 23756607
- [Background] Iwase S, Kawahara Y, Nishimura N, Sugenoya J. Effect of micro mist sauna bathing on thermoregulatory and circulatory functions and thermal sensation in humans. Int J Biometeorol. 2016 May;60(5):699-709. doi: 10.1007/s00484-015-1064-0. Epub 2015 Sep 18. PMID 26384686
- [Background] Jevtovic S, Karlovic D, Mihaljevic-Peles A, Seric V, Vrkic N, Jaksic N. Serum Brain-derived neurotrophic factor (BDNF): the severity and symptomatic dimensions of depression. Psychiatr Danub. 2011 Dec;23(4):363-9. PMID 22075737
- [Background] Ejiri J, Inoue N, Kobayashi S, Shiraki R, Otsui K, Honjo T, Takahashi M, Ohashi Y, Ichikawa S, Terashima M, Mori T, Awano K, Shinke T, Shite J, Hirata K, Yokozaki H, Kawashima S, Yokoyama M. Possible role of brain-derived neurotrophic factor in the pathogenesis of coronary artery disease. Circulation. 2005 Oct 4;112(14):2114-20. doi: 10.1161/CIRCULATIONAHA.104.476903. Epub 2005 Sep 26. PMID 16186425
- [Background] Katz A, Meiri N. Brain-derived neurotrophic factor is critically involved in thermal-experience-dependent developmental plasticity. J Neurosci. 2006 Apr 12;26(15):3899-907. doi: 10.1523/JNEUROSCI.0371-06.2006. PMID 16611805
- [Background] Kohara K, Kitamura A, Morishima M, Tsumoto T. Activity-dependent transfer of brain-derived neurotrophic factor to postsynaptic neurons. Science. 2001 Mar 23;291(5512):2419-23. doi: 10.1126/science.1057415. PMID 11264540
- [Background] Kojima D, Nakamura T, Banno M, Umemoto Y, Kinoshita T, Ishida Y, Tajima F. Head-out immersion in hot water increases serum BDNF in healthy males. Int J Hyperthermia. 2018 Sep;34(6):834-839. doi: 10.1080/02656736.2017.1394502. Epub 2017 Nov 20. PMID 29157042
- [Background] Kuennen M, Gillum T, Dokladny K, Bedrick E, Schneider S, Moseley P. Thermotolerance and heat acclimation may share a common mechanism in humans. Am J Physiol Regul Integr Comp Physiol. 2011 Aug;301(2):R524-33. doi: 10.1152/ajpregu.00039.2011. Epub 2011 May 25. PMID 21613575
- [Background] Kukkonen-Harjula K, Oja P, Laustiola K, Vuori I, Jolkkonen J, Siitonen S, Vapaatalo H. Haemodynamic and hormonal responses to heat exposure in a Finnish sauna bath. Eur J Appl Physiol Occup Physiol. 1989;58(5):543-50. doi: 10.1007/BF02330710. PMID 2759081
- [Background] Lang UE, Hellweg R, Gallinat J. BDNF serum concentrations in healthy volunteers are associated with depression-related personality traits. Neuropsychopharmacology. 2004 Apr;29(4):795-8. doi: 10.1038/sj.npp.1300382. PMID 14735133
- [Background] Laatikainen T, Salminen K, Kohvakka A, Pettersson J. Response of plasma endorphins, prolactin and catecholamines in women to intense heat in a sauna. Eur J Appl Physiol Occup Physiol. 1988;57(1):98-102. doi: 10.1007/BF00691246. PMID 2830109
- [Background] Laukkanen T, Khan H, Zaccardi F, Laukkanen JA. Association between sauna bathing and fatal cardiovascular and all-cause mortality events. JAMA Intern Med. 2015 Apr;175(4):542-8. doi: 10.1001/jamainternmed.2014.8187. PMID 25705824
- [Background] Laukkanen T, Kunutsor S, Kauhanen J, Laukkanen JA. Sauna bathing is inversely associated with dementia and Alzheimer's disease in middle-aged Finnish men. Age Ageing. 2017 Mar 1;46(2):245-249. doi: 10.1093/ageing/afw212. PMID 27932366
- [Background] Lasek-Bal A, Jedrzejowska-Szypulka H, Rozycka J, Bal W, Holecki M, Dulawa J, Lewin-Kowalik J. Low Concentration of BDNF in the Acute Phase of Ischemic Stroke as a Factor in Poor Prognosis in Terms of Functional Status of Patients. Med Sci Monit. 2015 Dec 14;21:3900-5. doi: 10.12659/msm.895358. PMID 26656843
- [Background] Lee E, Laukkanen T, Kunutsor SK, Khan H, Willeit P, Zaccardi F, Laukkanen JA. Sauna exposure leads to improved arterial compliance: Findings from a non-randomised experimental study. Eur J Prev Cardiol. 2018 Jan;25(2):130-138. doi: 10.1177/2047487317737629. Epub 2017 Oct 19. PMID 29048215
- [Background] Lee BJ, Miller A, James RS, Thake CD. Cross Acclimation between Heat and Hypoxia: Heat Acclimation Improves Cellular Tolerance and Exercise Performance in Acute Normobaric Hypoxia. Front Physiol. 2016 Mar 8;7:78. doi: 10.3389/fphys.2016.00078. eCollection 2016. PMID 27014080
- [Background] Leckie RL, Oberlin LE, Voss MW, Prakash RS, Szabo-Reed A, Chaddock-Heyman L, Phillips SM, Gothe NP, Mailey E, Vieira-Potter VJ, Martin SA, Pence BD, Lin M, Parasuraman R, Greenwood PM, Fryxell KJ, Woods JA, McAuley E, Kramer AF, Erickson KI. BDNF mediates improvements in executive function following a 1-year exercise intervention. Front Hum Neurosci. 2014 Dec 11;8:985. doi: 10.3389/fnhum.2014.00985. eCollection 2014. PMID 25566019
- [Background] Leppaluoto J, Huttunen P, Hirvonen J, Vaananen A, Tuominen M, Vuori J. Endocrine effects of repeated sauna bathing. Acta Physiol Scand. 1986 Nov;128(3):467-70. doi: 10.1111/j.1748-1716.1986.tb08000.x. PMID 3788622
- [Background] Leppaluoto J, Tuominen M, Vaananen A, Karpakka J, Vuori J. Some cardiovascular and metabolic effects of repeated sauna bathing. Acta Physiol Scand. 1986 Sep;128(1):77-81. doi: 10.1111/j.1748-1716.1986.tb07952.x. PMID 3766176
- [Background] Lewthwaite J, Owen N, Coates A, Henderson B, Steptoe A. Circulating human heat shock protein 60 in the plasma of British civil servants: relationship to physiological and psychosocial stress. Circulation. 2002 Jul 9;106(2):196-201. doi: 10.1161/01.cir.0000021121.26290.2c. PMID 12105158
- [Background] Lorenzo S, Halliwill JR, Sawka MN, Minson CT. Heat acclimation improves exercise performance. J Appl Physiol (1985). 2010 Oct;109(4):1140-7. doi: 10.1152/japplphysiol.00495.2010. Epub 2010 Aug 19. PMID 20724560
- [Background] Lorenzo S, Minson CT, Babb TG, Halliwill JR. Lactate threshold predicting time-trial performance: impact of heat and acclimation. J Appl Physiol (1985). 2011 Jul;111(1):221-7. doi: 10.1152/japplphysiol.00334.2011. Epub 2011 Apr 28. PMID 21527667
- [Background] Maass A, Duzel S, Brigadski T, Goerke M, Becke A, Sobieray U, Neumann K, Lovden M, Lindenberger U, Backman L, Braun-Dullaeus R, Ahrens D, Heinze HJ, Muller NG, Lessmann V, Sendtner M, Duzel E. Relationships of peripheral IGF-1, VEGF and BDNF levels to exercise-related changes in memory, hippocampal perfusion and volumes in older adults. Neuroimage. 2016 May 1;131:142-54. doi: 10.1016/j.neuroimage.2015.10.084. Epub 2015 Nov 3. PMID 26545456
- [Background] Masuda A, Koga Y, Hattanmaru M, Minagoe S, Tei C. The effects of repeated thermal therapy for patients with chronic pain. Psychother Psychosom. 2005;74(5):288-94. doi: 10.1159/000086319. PMID 16088266
- [Background] Matsuda N, Lu H, Fukata Y, Noritake J, Gao H, Mukherjee S, Nemoto T, Fukata M, Poo MM. Differential activity-dependent secretion of brain-derived neurotrophic factor from axon and dendrite. J Neurosci. 2009 Nov 11;29(45):14185-98. doi: 10.1523/JNEUROSCI.1863-09.2009. PMID 19906967
- [Background] Mero A, Tornberg J, Mantykoski M, Puurtinen R. Effects of far-infrared sauna bathing on recovery from strength and endurance training sessions in men. Springerplus. 2015 Jul 7;4:321. doi: 10.1186/s40064-015-1093-5. eCollection 2015. PMID 26180741
- [Background] Minson CT, Cotter JD. CrossTalk proposal: Heat acclimatization does improve performance in a cool condition. J Physiol. 2016 Jan 15;594(2):241-3. doi: 10.1113/JP270879. Epub 2015 Dec 14. PMID 26668072
- [Background] Moseley PL. Heat shock proteins and heat adaptation of the whole organism. J Appl Physiol (1985). 1997 Nov;83(5):1413-7. doi: 10.1152/jappl.1997.83.5.1413. PMID 9375300
- [Background] Morrison S, Sleivert GG, Cheung SS. Passive hyperthermia reduces voluntary activation and isometric force production. Eur J Appl Physiol. 2004 May;91(5-6):729-36. doi: 10.1007/s00421-004-1063-z. Epub 2004 Mar 11. PMID 15015001
- [Background] Molendijk ML, Haffmans JP, Bus BA, Spinhoven P, Penninx BW, Prickaerts J, Oude Voshaar RC, Elzinga BM. Serum BDNF concentrations show strong seasonal variation and correlations with the amount of ambient sunlight. PLoS One. 2012;7(11):e48046. doi: 10.1371/journal.pone.0048046. Epub 2012 Nov 2. PMID 23133609
- [Background] Morton JP, Kayani AC, McArdle A, Drust B. The exercise-induced stress response of skeletal muscle, with specific emphasis on humans. Sports Med. 2009;39(8):643-62. doi: 10.2165/00007256-200939080-00003. PMID 19769414
- [Background] Muller P, Rehfeld K, Schmicker M, Hokelmann A, Dordevic M, Lessmann V, Brigadski T, Kaufmann J, Muller NG. Evolution of Neuroplasticity in Response to Physical Activity in Old Age: The Case for Dancing. Front Aging Neurosci. 2017 Mar 14;9:56. doi: 10.3389/fnagi.2017.00056. eCollection 2017. PMID 28352225
- [Background] Nielsen B, Strange S, Christensen NJ, Warberg J, Saltin B. Acute and adaptive responses in humans to exercise in a warm, humid environment. Pflugers Arch. 1997 May;434(1):49-56. doi: 10.1007/s004240050361. PMID 9094255
- [Background] Nielsen B, Hales JR, Strange S, Christensen NJ, Warberg J, Saltin B. Human circulatory and thermoregulatory adaptations with heat acclimation and exercise in a hot, dry environment. J Physiol. 1993 Jan;460:467-85. doi: 10.1113/jphysiol.1993.sp019482. PMID 8487204
- [Background] Nybo L, Rasmussen P, Sawka MN. Performance in the heat-physiological factors of importance for hyperthermia-induced fatigue. Compr Physiol. 2014 Apr;4(2):657-89. doi: 10.1002/cphy.c130012. PMID 24715563
- [Background] Nybo L, Lundby C. CrossTalk opposing view: Heat acclimatization does not improve exercise performance in a cool condition. J Physiol. 2016 Jan 15;594(2):245-7. doi: 10.1113/JP270880. Epub 2015 Dec 14. No abstract available. PMID 26667955
- [Background] Pereira ES, Krause Neto W, Calefi AS, Georgetti M, Guerreiro L, Zocoler CAS, Gama EF. Significant Acute Response of Brain-Derived Neurotrophic Factor Following a Session of Extreme Conditioning Program Is Correlated With Volume of Specific Exercise Training in Trained Men. Front Physiol. 2018 Jul 3;9:823. doi: 10.3389/fphys.2018.00823. eCollection 2018. PMID 30018570
- [Background] Phillips C, Baktir MA, Das D, Lin B, Salehi A. The Link Between Physical Activity and Cognitive Dysfunction in Alzheimer Disease. Phys Ther. 2015 Jul;95(7):1046-60. doi: 10.2522/ptj.20140212. Epub 2015 Jan 8. PMID 25573757
- [Background] Rasmussen P, Brassard P, Adser H, Pedersen MV, Leick L, Hart E, Secher NH, Pedersen BK, Pilegaard H. Evidence for a release of brain-derived neurotrophic factor from the brain during exercise. Exp Physiol. 2009 Oct;94(10):1062-9. doi: 10.1113/expphysiol.2009.048512. Epub 2009 Aug 7. PMID 19666694
- [Background] Leak RK. Heat shock proteins in neurodegenerative disorders and aging. J Cell Commun Signal. 2014 Dec;8(4):293-310. doi: 10.1007/s12079-014-0243-9. Epub 2014 Sep 11. PMID 25208934
- [Background] Redberg RF. Health benefits of sauna bathing. JAMA Intern Med. 2015 Apr;175(4):548. doi: 10.1001/jamainternmed.2014.8206. No abstract available. PMID 25706401
- [Background] Rendell RA, Prout J, Costello JT, Massey HC, Tipton MJ, Young JS, Corbett J. Effects of 10 days of separate heat and hypoxic exposure on heat acclimation and temperate exercise performance. Am J Physiol Regul Integr Comp Physiol. 2017 Sep 1;313(3):R191-R201. doi: 10.1152/ajpregu.00103.2017. Epub 2017 Jun 7. PMID 28592459
- [Background] Sotiridis A, Debevec T, Mekjavic IB. Letter to the Editor: Combined effects of hypoxia and heat: importance of hypoxic dose. Am J Physiol Regul Integr Comp Physiol. 2018 Feb 1;314(2):R228-R229. doi: 10.1152/ajpregu.00347.2017. No abstract available. PMID 29388459
- [Background] Roberts CK, Vaziri ND, Barnard RJ. Effect of diet and exercise intervention on blood pressure, insulin, oxidative stress, and nitric oxide availability. Circulation. 2002 Nov 12;106(20):2530-2. doi: 10.1161/01.cir.0000040584.91836.0d. PMID 12427646
- [Background] Romeyke T, Scheuer HC, Stummer H. Fibromyalgia with severe forms of progression in a multidisciplinary therapy setting with emphasis on hyperthermia therapy--a prospective controlled study. Clin Interv Aging. 2014 Dec 19;10:69-79. doi: 10.2147/CIA.S74949. eCollection 2015. PMID 25565789
- [Background] Rothman SM, Mattson MP. Activity-dependent, stress-responsive BDNF signaling and the quest for optimal brain health and resilience throughout the lifespan. Neuroscience. 2013 Jun 3;239:228-40. doi: 10.1016/j.neuroscience.2012.10.014. Epub 2012 Oct 16. PMID 23079624
- [Background] Rudman D, Feller AG, Nagraj HS, Gergans GA, Lalitha PY, Goldberg AF, Schlenker RA, Cohn L, Rudman IW, Mattson DE. Effects of human growth hormone in men over 60 years old. N Engl J Med. 1990 Jul 5;323(1):1-6. doi: 10.1056/NEJM199007053230101. PMID 2355952
- See also: Brigadski T., and Leßmann V. BDNF: a regulator of learning and memory processes with clinical potential. e-Neuroforum 2014; 5, 1-11. doi: 10.1007/s13295- 014- 0053- 9 — https://link.springer.com/article/10.1007%2Fs13295-014-0053-9
- See also: Brenner I.K. et al. The impact of heat exposure and repeated exercise on circulating stress hormones. European Journal of Applied Physiology and Occupational Physiology.1997; 76(5): 445-454 — https://link.springer.com/article/10.1007/s004210050274
- See also: Brisson G., Boisvert P., Peronnet F., Quirion A., Senecal L. Face cooling-induced reduction of plasma prolactin response to exercise as part of an integrated response to thermal stress. Eur J Appl Physiol Occup Physiol 1989; 58: 816-820 — https://link.springer.com/article/10.1007%2FBF02332212
- See also: Campbell B., Zito G., Colquhoun R., Martinez N., St Louis C. et al. Inter- and intra-day test-retest reliability of the Cosmed FitmateProTM indirect calorimeter for resting metabolic rate. Kathryn Raines University of South Florida, Tampa, Florida, US — https://jissn.biomedcentral.com/articles/10.1186/1550-2783-11-S1-P46
- See also: Halcox Julian P.J., Deanfield John, Shamaei-Tousi Alireza, Henderson Brian, Steptoe Andrew, Coates Anthony R.M., Singhal Atul and Lucas Alan. Circulating Human Heat Shock Protein 60 in the Blood of Healthy Teenagers: A Novel Determinant of Endothelial — https://pdfs.semanticscholar.org/8755/0be8a1da4fd9cb342e66a79338451502bd15.pdf